CLINICAL TRIAL: NCT02100592
Title: Early Verticalization in neuroICU With ERIGO: a Safety and Feasibility Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERIGO-1
Record Dates: First submitted 2014-03-24; First posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Brain Injury
Keywords: brain injury; coma; intensive care; early rehabilitation
MeSH Terms: conditions — Brain Injuries; Coma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erigo treated (Experimental): Early rehabilitation treatment on Erigo Hocoma, a tilt table with integrated stepping device within 3 - 30 days from injury
  Interventions: Other: Early rehabilitation treatment on Erigo Hocoma

INTERVENTIONS:
Other: Early rehabilitation treatment on Erigo Hocoma — 5 weekly sessions of erigo for three weeks. Expected tilt angle up to 60 °
Other: Early rehabilitation treatment on Erigo Hocoma — Early verticalization treatment with Erigo Hocoma, a tilt table with stepping system

SUMMARY:
Severe brain injuries induce alteration of state of consciousness. These functional limitations can be significantly alleviated by treatment neurorehabilitation, particularly if this is established early. It has been shown that treatment of vertical integration in patients in a vegetative state or minimally conscious state can improve the level of supervision and positive influence on rehabilitation. Therefore, there are sufficient indications that anticipate the treatment of vertical integration, since the phase of hospitalization in ICUs, may improve the functional outcome of the patient.

DETAILED DESCRIPTION:
Early verticalization and stepping with the equipment Hocoma Erigo, during monitoring of vital parameters. The device Erigo is already CE marked and, for the purposes of the study, will be used in accordance with the intended use of the same mark (after-market clinical investigation).

ELIGIBILITY:
Inclusion Criteria:

1. Patient / a severe acquired brain injury occurred 3 to 30 days prior to enrollment
2. Age between 18 and 75 years
3. Glasgow Coma Scale ≤ 8 at entrance in ICUs
4. Adequate respiratory exchange with PaO2/FiO2 ≥ 250
5. Absence of sedation increased

Exclusion Criteria:

1. Major chest trauma with multiple rib fractures and / or pneumothorax
2. Presence of fractures, vascular lesions, skin lesions with loss of substance in the abdomen, pelvis or lower limb
3. Cardiovascular instability despite support with amines
4. Intracranial pressure (ICP)> 25 mm / Hg
5. Cerebral Perfusion Pressure (PPC) <60 mm / Hg
6. Severe kidney failure requiring replacement therapy
7. Decompensated liver disease
8. Hematocrit value of ≤ 30%
9. Body weight> 135 kg or height> 210 cm
10. Deep vein thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adverse events during verticalization | 21 days: from T1 (first session) to T15 (last session)
  It is a composite outcome, assessing the occurence of at least one of the following conditions (component outcomes):
  Heart rate <40 bpm or> 150 bpm; Mean arterial pressure <70 mmHg; Arterial oxygen saturation <90%; Onset of ECG anomalies; Traumatic dislodgement of a device;

SECONDARY OUTCOMES:
Changes of hemodynamic parameters | 21 days: from T1 (first session) to T15 (last session)
  Changes of hemodynamic parameters during each session and from T1 to T15; assessed parameters are:
  stroke volume; peripheral resistances; mean arterial pressure; cerebral perfusion pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Study Chair — Ospedale generale di zona 'Moriggia Pelascini'; Roberto Valsecchi, MD, Principal Investigator — Ospedale generale di zona 'Moriggia Pelascini'; Leopold Saltuari, MD, Principal Investigator — LDK Hochzirl; Luca Sebastianelli, MD, Principal Investigator — Ospedale generale di zona 'Moriggia Pelascini'